CLINICAL TRIAL: NCT03447444
Title: Dignity for Persons With Dementia and Signs of Frontotemporal Affection in Institutions.See us and Dance With us
Brief Title: Music and Physical Activity in Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Dagfinn Nåden, professor, Oslo Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Frontallob dementia
Record Dates: First submitted 2018-01-22; First posted 2018-02-27 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Dementia Frontal
Keywords: dignity; music therapy; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: case studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- music and physical activity (Other): An intervention consisting of physical activity, music and walking, was systematically implemented for eight weeks
  Interventions: Other: music and physical activity

INTERVENTIONS:
Other: music and physical activity — This feasibility study focus on promoting a combination of music therapy and physical activity with the primary goal to describe the influence on restlessness, irritability, and aggression in persons with severe stage of dementia with a mixture of symptoms including frontal lobe problems in institutional care. A secondary goal is to investigate the treatment fidelity.

SUMMARY:
Fronto lobe dementia constitutes 10-20 % of dementia conditions within younger persons (>65). People with neuronal degeneration in frontal and temporal lobes demonstrate a decline in social conduct, apathy, loss of insight that is gradual and progressive. Family members often experience guilt and shame because of the patients' behavior before institutionalization, and different behavioral disorders will cause great challenges to family caregivers and to staff after institutionalization. Preservation of dignity, both in regards to the person being affected, and their relatives, therefore seem highly relevant both before and after institutionalization.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate whether a combined intervention of physical activity and music therapy could reduce restlessness, irritability, and aggression among institutionalized people with severe dementia. An exploratory design was used to evaluate a combined intervention of physical activity, music therapy, and in- or outdoors walking daily, systematically implemented for eight weeks for persons with severe dementia in institutional care.

ELIGIBILITY:
Inclusion Criteria:Persons with dementia with symptoms of frontal lobe dementia, who had lived for at least 6 months in a unit special care dementia unit in a nursing home

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2015-02-27 (Actual); Study Completion 2015-02-27 (Actual)

PRIMARY OUTCOMES:
Brøset Violence Checklist | change from baseline to eight weeks into intervention
  The BVC assesses the presence of six observable patient behaviors, namely whether the patient is confused, irritable, boisterous, verbally threatening, physically threatening, and/or attacking objects

SECONDARY OUTCOMES:
Neuropsychiatric Inventory | baseline
  The Neuropsychiatric Inventory-Questionnaire [NPI-Q] is a clinical instrument for assessing behavioral and psychological symptoms in dementia

CONTACTS AND LOCATIONS:
Overall Officials: Dagfinn Nåden, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No